CLINICAL TRIAL: NCT05705479
Title: Shoulder Instability Trial Comparing Arthroscopic Stabilization Benefits Compared With Latarjet Procedure Evaluation
Brief Title: Shoulder Instability Trial Comparing Arthroscopic Stabilization Benefits Compared With Latarjet Procedure Evaluation - STABLE Definitive Trial
Acronym: STABLE-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Moin Khan, Associate Professor and Orthopaedic Surgeon, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STABLE-2
Record Dates: First submitted 2023-01-17; First posted 2023-01-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Dislocation; Sport Injuries; Anterior Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bankart + Remplissage Procedure (Experimental): Bankart Procedure: the participant will be placed in the lateral decubitus or beach chair position. Standard diagnostic arthroscopy will be performed. The anterior capsulolabral complex will be freed from the anterior aspect of the scapular neck. The anterior aspect of the scapular neck will be decorticated using a motorized burr. A capsuloligamentous repair will be performed with the capsule shifted from inferior to superior and repaired on the glenoid face. The number of anchors used for the repair will be left to the discretion of the surgeon. Patients will be given a sling for 4 weeks, and participation in sports will not be allowed for 6 months.
  Interventions: Procedure: Bankart + Remplissage Procedure
- Latarjet Procedure (Experimental): Open or Arthroscopic coracoid transfer (Latarjet Procedure): This procedure may be performed through small incisions (minimally invasive) but may require a larger incision in some cases. It involves the transfer of a nearby bony structure (the coracoid process) to the front of the shoulder joint (glenoid). This bone will then provide support to prevent the shoulder joint from dislocating.
  Interventions: Procedure: Latarjet Procedure

INTERVENTIONS:
Procedure: Bankart + Remplissage Procedure — Participants will undergo arthroscopic stabilization.
  Arms: Bankart + Remplissage Procedure
Procedure: Latarjet Procedure — Participants will undergo open or arthroscopic Latarjet procedure.
  Arms: Latarjet Procedure

SUMMARY:
The primary objective of the study is to evaluate the functional shoulder recovery of patients with recurrent shoulder dislocations at 24 months when treated with either arthroscopic capsuloligamentous repair (Bankart Procedure +/- Remplissage) or coracoid transfer (Latarjet procedure).

DETAILED DESCRIPTION:
Background:

Shoulder is a highly mobile joint with the most directional range of movement compared to other joints in the body. Thus, the surrounding supporting structures of the shoulder joint compromise on the stability of the joint, in order to accomplish this wide range of motion.

Anterior dislocations, the most common type of shoulder dislocation, are often complicated by instability, and repeated dislocations. Shoulder instability results in pain and negatively impacts quality of life. Several long-term studies have demonstrated a relationship between the repeated dislocations and the risk of arthritis.

Surgical stabilization of the shoulder improves function and may reduce the risk of developing degenerative arthritis. Two procedures are commonly performed in patients with repeated dislocations: a bony transfer procedure (Latarjet) or a soft tissue procedure (Bankart + Remplissage). The Latarjet procedure involves transferring bone to the front of the shoulder. The Bankart + Remplissage procedure involves tightening the soft tissues at the front of the shoulder joint.

Although retrospective clinical studies have suggested a reduced recurrence rate with the Latarjet procedure, there is a higher reported complication rate and potential morbidity associated with the open procedure. Several case series from high-volume surgeons in Europe have suggested the Latarjet repair to be an acceptable and potentially favorable surgical approach for all cases of recurrent anterior shoulder dislocation, even in the primary setting and in the absence of significant glenoid cup bone loss. Retrospective analysis of soft tissue repair in comparison to open coracoid (Latarjet) procedure found at 10-year follow up, redislocation rates were 13% (36) of 271 shoulders with a Bankart repair and 1% (1) of the 93 shoulders with a Latarjet repair.

Need for a Pilot Study Prior to a Large Trial:

No comparative randomized control trial has been completed evaluating Bankart repair in comparison to Latarjet procedure in the setting of mild to moderate bone loss. Thus, surgeons face uncertainty regarding which procedure to perform. The Latarjet is more invasive (larger incision) and some research suggests it may be more effective at treating instability. The Bankart procedure, while minimally invasive (smaller incision), may result in higher rates of instability after surgery.

Study Aims and Objectives:

The primary objective of the study is to evaluate the functional shoulder recovery of patients with recurrent shoulder dislocations at 24 months when treated with either arthroscopic capsuloligamentous repair (Bankart Procedure +/- Remplissage) or coracoid transfer (Latarjet procedure).

Our trial will compare arthroscopic capsuloligamentous repair vs. coracoid transfer (Latarjet procedure) on:

1. Rates of recurrent shoulder dislocations and symptoms of instability up to 24 months' post- surgery;
2. Clinical outcomes measured by American Shoulder and Elbow Society (ASES) score, Shoulder Activity Scale and EQ-5D and Patient Satisfaction Scale;
3. Physical examination: range of motion, strength, stability;
4. Return to previous level of activity;
5. Rate of shoulder-related complications and serious adverse events.

Study Design:

The investigators propose a multi-center pilot Randomized Clinical Trial of 126 patients across Canada, United States, Chile and Europe to compare the effect of capsuloligamentous repair (Bankart + Remplissage procedure) and coracoid transfer (Latarjet procedure) in patients with post-traumatic recurrent anterior dislocation. Eligible and consenting participants will be followed-up by the site for 24 months. Outcomes will be assessed at 2 weeks, 3 months, 6 months, 12 months, and 24 months post-surgery. Eligible participants will be randomized to one of two treatment groups:

Arthroscopic capsuloligamentous repair (Bankart + Remplissage Procedure) Open or Arthroscopic coracoid transfer (Latarjet Procedure) Once participants have provided informed consent, baseline demographics, relevant medical history, and details regarding their diagnosis will be collected from the participant, the attending surgeon, their medical record and through physical examination. Participants will also complete The Western Ontario Shoulder Instability Index (WOSI) and he American Shoulder and Elbow Surgeons questionnaire (ASES) at the time of enrolment.

After surgery, surgical and peri-operative details will be collected from the attending surgeon and the participant's medical records. Adverse events occurring during the surgical procedure or perioperative period will also be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-50 years;
2. Diagnosis of post-traumatic recurrent anterior dislocation. This will require a minimum of 2 episodes of documented dislocations either by radiographic evidence or documented reduction of anterior shoulder dislocation as well as physical examination eliciting unwanted glenohumeral translation with reproduction of symptoms;
3. Subcritical glenoid bone loss as defined on CT by standardized and reproducible best-fit circle technique (>10% but <20%);
4. Provision of informed consent.

Exclusion Criteria:

1. Patients with concomitant injuries of the index shoulder (cuff tear, greater tuberosity fracture);
2. Previous shoulder surgery;
3. Patients that will likely have problems, in the judgment of the investigators, with maintaining follow-up;
4. Epilepsy/seizure disorder;
5. Patients who are currently incarcerated;
6. Diagnosis of multidirectional instability;
7. Cases involving litigation or workplace insurance claims (e.g. WSIB);
8. Confirmed connective tissue disorder (Ehlers-Danlos, Marfans) or Beighton hypermobility score > 6.
9. Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome - Shoulder function | 2 years
  The change from baseline to 24 months post-intervention difference in Western Ontario Shoulder Instability Index (WOSI) scores between patients with recurrent dislocations treated with Bankart Procedure + Remplissage versus Latarjet procedure.

SECONDARY OUTCOMES:
Rate of Recurrence | 2 years
  Rate of recurrent dislocation and symptomatic instability between patients randomized to (capsuloligamentous repair + remplissage) and those receiving open Latarjet procedure.
Clinical Outcome | 2 years
  Measured by ASES questionnaire (American Shoulder and Elbow Surgeons)
Clinical Outcome - Quality of Life | 2 years
  Measured by EQ-5D
Clinical Outcome - Shoulder activity | 2 years
  Measured by Shoulder Activity Scale
Rate of participants with anterior shoulder instability | 2 years
  Measured by apprehension-relocation physical examination maneuver
Rate of participants with full range of motion | 2 years
  Assessed in forward flexion, abduction, external rotation and internal rotation.
Rate of participants that return to previous level of activity | 2 years
  Return to previous level of activity and sport (self reported)
Rate of major and minor shoulder-related complications and serious adverse events | 2 years
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan M, Bedi A, Degen R, Warner J, Bhandari M; STABLE Investigators. Multicentre randomised controlled trial comparing Bankart repair with remplissage and Latarjet procedure in shoulder instability with subcritical bone loss (STABLE): study protocol. BMJ Open. 2024 Nov 14;14(11):e089831. doi: 10.1136/bmjopen-2024-089831. PMID 39542469